CLINICAL TRIAL: NCT03768804
Title: Assessing the Effect of the SyncAV Algorithm in Cardiac Resynchronization Therapy on Exercise Capacity and QRS Duration on Exercise
Brief Title: SyncAV Study: Investigation of the Efficacy of the SyncAV Fusion Pacing Algorithm on Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13808
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure, Systolic
Keywords: Cardiac resynchronisation therapy; Fusion pacing; SyncAV
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Intervention Model Description: Double blind, randomised crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SyncAV algorithm on (Other): Device randomised to have SyncAV on, with delta programmed to the value which gives the narrowest QRS duration at rest and pseudo left ventricular ("LV") only pacing
  Interventions: Other: SyncAV algorithm on
- SyncAV algorithm off (Other): Device randomised to have SyncAV off, with a fixed sensed atrioventricular ("AV") delay of 120ms or shorter if necessary to prevent fusion, and biventricular ("BiV") pacing
  Interventions: Other: SyncAV algorithm off

INTERVENTIONS:
Other: SyncAV algorithm on — Cardiac Resynchronisation Device will be set to have the SyncAV algorithm on for the duration of the cardiopulmonary exercise test ("CPET"), before being reset to pre-existing settings
  Arms: SyncAV algorithm on
Other: SyncAV algorithm off — ardiac Resynchronisation Device will be set to have the SyncAV algorithm off and a fixed AV delay, for the duration of the CPET, before being reset to pre-existing settings
  Arms: SyncAV algorithm off

SUMMARY:
In patients with weak pumping function of the heart, uncoordinated contraction of the chambers can be corrected using a cardiac resynchronization therapy ("CRT") pacemaker. These devices make patients live longer by improving how the heart pumps and reducing symptoms such as breathlessness. However, not all patients benefit from CRT and programming devices optimally can greatly influence success. Predicting the correct timings of contraction between the atria (top chambers of the heart) and the ventricles (bottom chambers), as well as between the left and right ventricles, especially when heart rate increases during exercises, is challenging.

A new approach to optimizing CRT programming has been proposed known as 'fusion-pacing'. This allows the electrical wave from the heart's own conduction system to merge or fuse with the impulse from the pacemaker in the left ventricle. The timing of the pacemaker's impulse is continuously adjusted to measurements the device makes of the hearts natural conduction. What is not clear is how effective 'fusion-pacing' is during exercise when the hearts natural conduction changes rapidly and unpredictably. We plan to investigate this by monitoring the electrocardiogram ("ECG") whilst accurately measuring exercise performance and ability during a cardiopulmonary exercise test ("CPET") on an exercise bike. We will also ask participants to rate their perceived exercise intensity to see whether fusion pacing improves ECG resynchronization, exercise performance, and patients' symptoms compared to standard programming.

DETAILED DESCRIPTION:
Heart failure represents a significant health problem, with the last national heart failure audit demonstrating prevalence in the United Kingdom of 900,000 patients, accounting for 5% of all acute hospital admissions. This is expected to increase with an ageing population. Despite improvements in medical therapy, prognosis remains poor, with an in- hospital mortality of 9.6%, and an estimated mortality of 30-40% at 1 year after diagnosis.

Multiple randomised controlled trials have demonstrated that cardiac resynchronization therapy pacemaker devices ("CRT") are an effective therapy for patients with poor pumping function and altered electrical conduction of the heart (left bundle branch block, "LBBB"), improving both morbidity and mortality. However, only 60-70% of patients notice a symptomatic improvement with CRT and even in patients who do respond, response can often be improved further by optimising how the device is programmed.

CRT devices improve coordination of heart pumping by pacing both ventricles of the heart. A key function of this is to coordinate the timing of contraction of the the atria and the ventricles (atrio-ventricular, or "AV", optimisation). This allows maximal filling of the left ventricle with blood. More recently, it has become important not only in standard bi-ventricular ("BiV") pacing, but to allow left ventricular pacing to be timed with intrinsic conduction to the right ventricle to provide CRT (so called 'fusion' pacing).

Multiple methods have been described to assess AV optimisation, including echocardiographic measurements. However, echo based methods are labour intensive, and their value is uncertain. Device algorithms utilising analysis of the intra-cardiac electrogram ("IEGM") have become an attractive alternative due to their rapid and automated nature, although evidence suggests that they may not have clinical benefit over using fixed AV delays. In addition, intrinsic AV conduction is known to alter with exercise, normally becoming shorter. Optimisation of AV delays in CRT on exercise has been shown to improve cardiac output. Device algorithms can therefore allow dynamic adjustment of AV delays as they change with exercise and heart rate (rate-adaptive AV delay or "RAAVD"). Indeed, use of individually tailored RAAVD in CRT patients has demonstrated an increase in exercise capacity.

Patients with heart failure and LBBB often have normal intrinsic right ventricular activation through the right bundle. Utilization of timed left ventricular ("LV") pacing to merge (or fuse) with this intrinsic conduction may confer benefits over standard BiV pacing, but requires relatively normal intrinsic AV conduction as well as correct timing of LV pacing to right ventricular ("RV") activation. Algorithms now exist which allow dynamic reassessment of intrinsic conduction and so adjustment of the optimal AV delay. They can therefore compensate for changes in the intrinsic AV delay on exercising, and so maintain adequate fusion pacing and CRT optimisation. One such software algorithm is SyncAV, developed by Abbott (Abbott Vascular, 3200 Lakeside Drive, Santa Clara, California 95054-2807). SyncAVTM assesses intrinsic AV conduction every 256 beats. It then sets a shorter programmed AV delay by subtracting a set period (known as the "delta" - adjustable but nominally set to 50ms) from the intrinsic time.

There is some evidence that fusion pacing gives benefit in terms of both acute pumping function of the heart and long term response to CRT. However, what remains unclear is whether the effect of dynamic AV optimisation and fusion pacing is maintained on exercise. Firstly, the re-analysis and adjustment intervals may be insufficient to allow effective fusion throughout exercise. It is therefore possible that with rapidly changing heart rates this coordinated timing is lost, leading to inefficient conduction of electricity through the heart. This could result in large periods of time on exercising without effective CRT and so poor exercise tolerance. Secondly, there is evidence that in patients with heart failure AV intervals do not alter with change in heart rate in a similar way to healthy controls. One study found that the degree of change is greater on exercise, whilst one demonstrated that in a CRT population only a third of patients had shorter optimal AV delay intervals on exercise, with a third being unchanged and a third longer. The use of a fixed "delta" in SyncAVTM may therefore result in incorrect adjustment of AV intervals as intrinsic conduction changes, with the effectiveness of SyncAV therefore depending on how the intrinsic interval changes.

We will use a prospective single-centre randomized single-blind crossover study to investigate the effectiveness of SyncAV on exercise, by randomising participants to either use of SyncAV or fixed AV delays, and then carrying out cardiopulmonary exercise testing ("CPET").

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and able to give informed consent.
* Patients with existing cardiac resynchronization therapy ("CRT") devices able to utilise the SyncAV algorithm, implanted ≥6 months and under follow up at Oxford University Hospitals National Health Service ("NHS") Foundation Trust.
* Evidence of response to CRT, defined as functional improvement or left ventricular ("LV") remodelling on imaging.
* Sinus rhythm and PR interval <250ms.
* Able to exercise to perform cardiopulmonary exercise testing ("CPET").

Exclusion Criteria:

* Pregnancy or breast feeding.
* Atrial fibrillation or atrial tachycardia.
* Underlying 2nd or 3rd degree heart block.
* PR interval ≥250ms.
* Chronotropic incompetence, defined as use of rate-response algorithm or ≥80% atrial pacing.
* Any concurrent condition contraindicating use of CPET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 1 Year
  Exercise capacity as measured by cardiopulmonary exercise testing ("CPET") including blood sampling
BORG-RPE rating | 1 Year
  Borg rating of perceived exertion ("Borg-RPE") during CPET

SECONDARY OUTCOMES:
QRS duration | 1 Year
  QRS duration during exercise, compared to at rest
Exercise duration | 1 Year
  Exercise duration as measured by cardiopulmonary exercise testing ("CPET")
PR duration | 1 Year
  Intrinsic PR duration during exercise when fusion pacing is on

CONTACTS AND LOCATIONS:
Overall Officials: Neil Herring, BMBCh MRCP, Principal Investigator — University of Oxford
Locations (1):
- Department of Physiology, Anatomy and Genetics, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD to be shared